CLINICAL TRIAL: NCT01488292
Title: Multi-Component Mental Health & Academic Intervention for Student Reintegration
Brief Title: RECAP Multi-Component Intervention Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan Han, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090633; R01MH077596 (NIH)
Record Dates: First submitted 2011-11-23; First posted 2011-12-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2014-12

CONDITIONS: Behavioral Problems; Emotional Problems
Keywords: mental health; social skills
MeSH Terms: conditions — Problem Behavior; Psychological Well-Being; Social Skills

ARMS (2):
- RECAP social skills and reading program (Experimental)
  Interventions: Behavioral: RECAP social skills and reading program
- Control group (services as usual) (No Intervention): Control Group (services as usual)

INTERVENTIONS:
Behavioral: RECAP social skills and reading program — weekly individual and group sessions
  Arms: RECAP social skills and reading program

SUMMARY:
This study evaluates the efficacy of the RECAP Mental Health + Academic Program for special education students in behavioral classrooms. The program includes multiple service components: the RECAP classroom mental health curriculum, which develops students' behavioral and social skills; reading intervention; individualized skills training; and parent group. Schools are randomly assigned to the treatment or control group. This two-year multi-component mental health and academic intervention is hypothesized to improve students' mental health, social skills, and academic functioning.

DETAILED DESCRIPTION:
Background Information

This research project evaluates the efficacy of the RECAP Mental Health + Academic Program, a two-year multi-component intervention for special education students in behavioral classrooms. The program has been shown to reduce students' emotional and behavioral problems and remediate academic deficits, particularly with regard to reading skills, in order to enhance academic and behavioral functioning and to facilitate special education students' appropriate transition and reintegration into the mainstream educational setting.

Using an educational and instructional approach that is familiar to school staff and students, RECAP helps teachers and parents to assist children in the development of behavioral and emotional skills that facilitate children's ability to learn and to solve problems adaptively. Many of the techniques and strategies used in RECAP are familiar to teachers, as RECAP represents an integration of basic behavioral principles. Its unique strength lies in its consistent and integrated framework, which provides a common language for students, teachers, and parents to talk about behavioral expectations and positive skills for children to learn and apply in everyday situations. Moreover, the RECAP program focuses on helping students resolve the behavioral and emotional problems that interfere with their own learning as well as the learning of other students in the classroom (e.g., due to lost instructional time via classroom disruption). In addition to this mental health curriculum, the intervention includes a reading intervention component that has been shown to significantly improve the academic progress of students with emotional and behavioral problems. In addition to the obvious fundamental need for direct remediation of this academic skills deficit that is common among these students, the reading intervention is designed to prepare special education students to participate in the academic instruction of the general education classroom at a functionally adaptive level.

Participating schools are randomly assigned to either receive the RECAP program or serve as a comparison school (services as usual). Student outcomes will be evaluated in the fall and spring of two school years, using behavioral observation, academic testing, and teacher-, parent-, and child-reports of psychopathology and social skills.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in behavioral classroom

Exclusion Criteria:

* Lack of legal guardian to provide consent

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2009-08; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in child emotional and behavioral problems | Baseline & 18 months
  Teacher TRF, Parent CBCL, Student SBQ ratings
Change in Woodcock Reading Mastery Test | Baseline & 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Han, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States